CLINICAL TRIAL: NCT03809689
Title: Study of Acute and Chronic Myocardiac Lesions Angiogenesis by 68Ga-NODAGA-RGD Cardiac PET
Brief Title: Study of Cardiac Lesions Angiogenesis by 68Ga-NODAGA-RGD Cardiac PET
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, PhD, MD, Head of Nuclear Medicine Department, University of Lausanne Hospitals
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-NODAGA-RGD cardiac PET
Record Dates: First submitted 2018-12-02; First posted 2019-01-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Myocardial Infarction, Acute; Myocardial Reperfusion; Chronic Ischemic Heart Disease
Keywords: Acute myocardial infarction; Myocardial reperfusion treatment; Chronic ischemic occlusion; 68Ga-NODAGA-RGD
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- acute infarction (Other): patients will have a 82-Rb and a 68Ga-NODAGA-RGD PET/CT at 1, 4 and 12 weeks after cardiac event
  Interventions: Other: 68Ga-NODAGA-RGD PET/CT; Diagnostic Test: 82-Rb PET/CT as part of standard care, not a comparator
- acute infarction requiring reperfusion (Other): patients will have a 82-Rb and a 68Ga-NODAGA-RGD PET/CT at 1, 4 and 12 weeks after cardiac event
  Interventions: Other: 68Ga-NODAGA-RGD PET/CT; Diagnostic Test: 82-Rb PET/CT as part of standard care, not a comparator
- chronic ischemic occlusion (Other): patients will have a 82-Rb and a 68Ga-NODAGA-RGD PET/CT before and 2 months after reperfusion treatment
  Interventions: Other: 68Ga-NODAGA-RGD PET/CT; Diagnostic Test: 82-Rb PET/CT as part of standard care, not a comparator

INTERVENTIONS:
Other: 68Ga-NODAGA-RGD PET/CT — intravenous injection of 200 Megabecquerel (MBq) 68Ga-NODAGA-RGD followed by a whole-body acquisition after injection and one hour after injection
Diagnostic Test: 82-Rb PET/CT as part of standard care, not a comparator — 2 intravenous injections of standard dose of 82-Rb : the first followed by an at-rest acquisition, the second followed by a pharmacological myocardial stress acquisition

SUMMARY:
The study is about exploring physiological angiogenesis linked to tissue repair in patients with acute heart infarction or chronic heart ischemia by means of 68Ga-NODAGA-RGD PET/CT imaging.

DETAILED DESCRIPTION:
Several animal studies have demonstrated the expression of αvβ3 integrins on the surface of the endothelium present in neovessels in formation, especially during neoangiogenesis after myocardial ischemic injury.

68Ga-NODAGA-RGD is a positron-emission-tomography (PET) ligand targeted towards αvβ3 integrins. αvβ3 integrins could potentially act as a biomarker for the follow-up of heart infarction.

In the present study, 68Ga-NODAGA-RGD PET/CT imaging is a tool to understand and evaluate tissue repair after heart lesion and its evolution allowing a better management of patients with occluded artery.

Three groups of patients are included : patients with acute infarction, patients with acute infarction requiring reperfusion treatment and patients with chronic ischemic occlusion.

Each patient would benefit from a 82Rb (82rubidium) PET/CT as part of standard management and from a 68Ga-NODAGA-RGD PET/CT as part of the present study.

Patients from groups 1 and 2 will have 3 sets of both exams : one after the ischemic event, one at one month and another at 3 months post event.

Patients form group 3 will have a set of both exams before reperfusion treatment and one at 2 months after reperfusion.

ELIGIBILITY:
Inclusion Criteria:

* patients with acute infarction or patients with acute infarction requiring reperfusion treatment or patients with chronic ischemic occlusion
* Karnofsky ≥ 80%
* signed informed consent

Exclusion Criteria:

* pregnancy, breastfeeding
* claustrophobia
* contra-indication to adenosine administration
* lack of discernment to sign informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
82Rb PET/CT : assessment of change of myocardial blood flow at rest and at stress | at 1, 4 and 12 weeks post ischemic events for patients of groups 1 and 2 - Before and 2 months after reperfusion treatment for patients of group 3
  mL/min/g
82Rb PET/CT : assessment of change of myocardial blood flow reserve at rest and at stress | at 1, 4 and 12 weeks post ischemic events for patients of groups 1 and 2 - Before and 2 months after reperfusion treatment for patients of group 3
  mL/min/g
82Rb PET/CT : assessment of change of difference of myocardial blood flow at stress and at rest | at 1, 4 and 12 weeks post ischemic events for patients of groups 1 and 2 - Before and 2 months after reperfusion treatment for patients of group 3
  mL/min/g
68Ga-NODAGA PET/CT : assessment of change of standard uptake value (SUV) | at 1, 4 and 12 weeks post ischemic events for patients of groups 1 and 2 - Before and 2 months after reperfusion treatment for patients of group 3
  g/ml

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, PhD, MD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No